CLINICAL TRIAL: NCT04019938
Title: Association of Cystatin C and Bone Mineral Density in Diabetic Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, XiaoChun Shu, Chief Physician, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZDWY(2019) K12-1
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal; Diabetes Mellitus
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Diabetes Mellitus | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Diabetic adults
  Interventions: Radiation: Dual-energy X-ray absorptiometry

INTERVENTIONS:
Radiation: Dual-energy X-ray absorptiometry — Cystatin C is measured as a part of routine investigation at the time of admission.

SUMMARY:
Type 1 diabetes is associated with low bone mineral density(BMD) and type 2 diabetes with normal or high BMD.

Cystatin C is a small molecule that is used to measure kidney function but it's not a troponin of the kidney. It has been associated with many other diseases like atrial fibrillation, depressive symptoms, melanoma, etc.

This crossectional clinical study was done to evaluate the association between Cystatin C and Bone mineral density in both types of diabetic patients.

DETAILED DESCRIPTION:
This is a cross-sectional study of adults with diabetes to determine the association of cystatin C with bone mineral density(BMD). All the inpatient in the department of endocrinology and metabolism in the fifth affiliated hospital of Sun Yat-Sen University will be screened for 5 to 6 months. Those satisfying the inclusion and exclusion criteria will be included in the study after signing the informed consent.

The patient's blood will be withdrawn in the morning after 8 hours of fasting and sent to the laboratory of the hospital for blood lipids, Hba1c, urinary Albumin creatinine ratio, uric acid, GGT, vitamin D, calcium, cystatin C, βserum collagen type 1 cross-linked C-telopeptide(βCTX),procollagen type I N-terminal propeptide( P1NP), phosphorus, alkaline phosphatase. Smoking habits, duration of diabetes, diabetes medications, and fracture history will be asked. The history of smoking is classified as

1. Non-smokers: Subjects who have never smoked any products (cigarettes, pipes or cigars) during their lifetime;
2. Smoking cessation: a person who smokes one or more products but stops smoking at least one month prior to the baseline survey;
3. Current smokers: A subject or any other product that smokes at least one cigarette per day.

The pelvic BMD, Vertebral body BMD will be measured in the physical examination department of the hospital and divided into normal, osteopenia, osteoporosis.

All covariates will be extracted to SPSS v.23 for statistical analysis to evaluate the association of Cystatin C and BMD.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes male / female, older than 50 years old.

Exclusion Criteria:

* Use of any drug that affects bone metabolism (bisphosphonate, denosumab, teriparatide, steroids, anticancer drugs, thyroid hormones, antidepressants, antiretrovirals, calcium, vitamins A/D)
* Any disease affecting bone minerals (hyperthyroidism, hypothyroidism, parathyroid disease, Cushing's disease, rickets/osteomalacia, collagen disorders, rheumatoid arthritis)
* Kidney disease, urinary albumin-creatinine ratio greater than 30 mg / g or GFR <60ml / min / 1.73m2.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient in the department of endocrinology and metabolism in the fifth affiliated hospital of Sun Yat-Sen University.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-12-25 (Estimated); Study Completion 2019-12-25 (Estimated)

PRIMARY OUTCOMES:
Serum Cystatin C | 6 months
  It is measured as a part of routine investigation at the time of admission

SECONDARY OUTCOMES:
Bone mineral density | 6 months
  Bone mineral density is measured using the Dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chun Shu, Principal Investigator — Fifth affiliated hospital of Sun Yat-Sen University; Ashish Shrestha, Principal Investigator — Fifth affiliated hospital of Sun Yat-Sen University
Locations (1):
- Ashish Shrestha, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No